CLINICAL TRIAL: NCT00656656
Title: Combined Treatment of Autoimmune Bullous Diseases With Protein A Immunoadsorption, Dexamethasone Pulse Therapy and Rituximab
Brief Title: Immunoadsorption, Dexamethasone Pulse Therapy and Rituximab for Pemphigus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Michael Kasperkiewicz, Dermatologist, University of Luebeck
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pemphigus-Luebeck
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Results first posted 2016-12-22 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-01

CONDITIONS: Pemphigus
Keywords: pemphigus; rituximab; immunoadsorption; dexamethasone; treatment; management
MeSH Terms: conditions — Pemphigus | interventions — Rituximab; Dexamethasone; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Immunoadsorption/Dexamethasone/Rituximab (Other)
  Interventions: Drug: Combination of Protein A Immunoadsorption, Rituximab, Dexamethasone plus Azathioprine

INTERVENTIONS:
Drug: Combination of Protein A Immunoadsorption, Rituximab, Dexamethasone plus Azathioprine — Protein A Immunoadsorption: performed on 3 consecutive days every 3 weeks
  Rituximab: 1000 mg i.v. given twice at a 2-week interval
  Dexamethasone pulse therapy: 100 mg i.v. given on 3 consecutive days every 3 weeks
  Azathioprine: 2.5 mg/kg body weight daily p.o.

SUMMARY:
Pemphigus is a severe autoimmune blistering disease mediated by circulating antibodies against certain proteins important for maintaining skin integrity. Protein A immunoadsorption is a dialysis-like technique selectively removing the antibodies from patient's blood. Rituximab is a synthetic antibody capable of destroying B cells. B cells are responsible for production of antibodies in the patients blood that, in turn, lead to clinical signs of pemphigus. Dexamethasone pulse therapy is a high-dose short-term corticosteroid therapy that may be used to suppress autoantibody production in pemphigus. While each of these three therapies had been used to treat pemphigus, none was shown effective in all cases. The hypothesis of this study is that a combination of protein A immunoadsorption, rituximab and dexamethasone is more effective that either of these treatments alone in achieving a rapid and durable improvement or cure in patients with pemphigus.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pemphigus confirmed by immunofluorescence and desmoglein ELISA.
* Severe disease or past treatment(s) not effective or past treatment(s) not tolerated.

Exclusion Criteria:

* General condition too poor to tolerate immunoadsorption treatment.
* Severe dementia or psychiatric disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Detlef Zillikens, MD, Principal Investigator — Department of Dermatology, University of Luebeck
Locations (1):
- Department of Dermatology, University of Luebeck, Lübeck, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Immunoadsorption/Dexamethasone/Rituximab: Combination of Protein A Immunoadsorption, Rituximab, Dexamethasone plus Azathioprine/Mycophenolate mofetil
  Protein A Immunoadsorption: performed on 3 consecutive days every 3-4 weeks
  Rituximab: 1000 mg i.v. given twice at a 2-week interval
  Dexamethasone pulse therapy: 100 mg i.v. given on 3 consecutive days initially every 3 weeks
  Azathioprine: 2.5 mg/kg body weight daily p.o.
  Mycophenolate mofetil 2 g/d p.o.
Period: Overall Study
Arm/Group | Immunoadsorption/Dexamethasone/Rituximab
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Immunoadsorption/Dexamethasone/Rituximab
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 6
Age, Continuous [Mean (Full Range); unit: years] | 55 [26 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 12
Region of Enrollment [Number; unit: participants]
  Germany | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving a Short- and Long-term Remission of Pemphigus
Description: Clinical remission was graded as partial remission on therapy, complete remission on therapy and complete remission off therapy, as described by Murell et al, J Am Acad Dermatol, 2008; 58:1043-6.
Time Frame: up to 43 months
Measure: Count of Participants; unit: Participants
Arm/Group | Immunoadsorption/Dexamethasone/Rituximab
Number analyzed (Participants) | 23
Participants | 23

2. Secondary Outcome: Number of Patients Who Experienced Side-effects of Treatment
Description: Patients who experienced side-effects were counted. In addition, the nature and severity of side-effects were recorded.
Time Frame: up to 43 months
Measure: Count of Participants; unit: Participants
Arm/Group | Immunoadsorption/Dexamethasone/Rituximab
Number analyzed (Participants) | 23
Participants | 2

ADVERSE EVENTS:
Arm/Group | Immunoadsorption/Dexamethasone/Rituximab
Serious Adverse Events (participants affected / at risk) | 2/23
Other Adverse Events (participants affected / at risk) | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Immunoadsorption/Dexamethasone/Rituximab (N=23)
Sepsis (Infections and infestations) | 1
extensive herpes simplex (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes